CLINICAL TRIAL: NCT03883932
Title: Fatherhood Focused Family Violence Education Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2000022823
Record Dates: First submitted 2019-03-18; First posted 2019-03-21 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Domestic Violence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- F3 Program (Experimental): The F3 group will focus on the fatherhood role each session. The topic of children and parenting will be applied to each of the standard FVEP topics.
  Interventions: Behavioral: Fatherhood Focused FVEP (F3)
- FVEP Program (Active Comparator): A retrospective control group who received the standard FVEP will be included in this arm.
  Interventions: Behavioral: Family Violence Education Program (FVEP)

INTERVENTIONS:
Behavioral: Fatherhood Focused FVEP (F3) — F3 is designed to focus specifically on the importance of fathering within a cognitive-behavioral intervention.
  Arms: F3 Program
Behavioral: Family Violence Education Program (FVEP) — FVEP is a court-mandated program intended to treat those arrested for intimate partner violence (IPV).
  Arms: FVEP Program

SUMMARY:
The purpose of this study is to explore the feasibility of a novel intervention approach for fathers arrested for an initial episode of intimate partner violence (IPV) by systematically developing an alternate version of a standard, statewide, court-mandated Family Violence Education Program (FVEP) to focus specifically on the importance of fathering within a cognitive-behavioral intervention to be called Fatherhood Focused FVEP (F3).

DETAILED DESCRIPTION:
This study will aim to modify the treatment as usual FVEP framework to be father focused. Materials will be developed to accommodate the change in scope of program focus for the purposes of training and supervising group leaders. An evaluation of the fidelity to the original FVEP model will be assessed through the review of service delivery.

In addition, the acceptability of Fatherhood Focused FVEP (F3) will be compared to the treatment as usual, FVEP as it is presently implemented. To do this, fathers who participate in FVEP will be compared to men who participate in F3 around the constructs: group cohesion, motivation to change, satisfaction with the program and rates of successful completion. Tertiary outcomes will include the assessment of: aggression toward intimate partners and hostile-aggressive parenting behaviors as reported on assessment measures and subsequent arrest records.

ELIGIBILITY:
Inclusion Criteria:

* Fathers referred to the FVEP program as a pretrial diversion following their first arrest for an incident of IPV with a female partner.
* Fathers must have at least one biological child under the age of 18.
* Fathers must have at least monthly contact with one of their biological children.

Exclusion Criteria:

* Fathers will be excluded if they are arrested for violence perpetrated against someone other than a current or former female partner.
* Fathers will be excluded if there is evidence of psychotic of suicidal symptoms on the Brief Symptom Inventory.
* Fathers will be excluded if they unable to complete questionnaires and group intervention in English.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2021-02-11 (Actual)

PRIMARY OUTCOMES:
Recidivism Incidence | 12 Months
  Recidivism will be determined through the review of state arrest records for additional IPV arrests.

SECONDARY OUTCOMES:
Group Cohesion | 3, 6 and 9 weeks
  Group cohesion will be assessed using Group Attitude Scale. Group Attitude scale is a self report instrument that consists of 20 items. The range of scores is from 20 to 180, where a higher score indicates WORSE cohesion.
Motivation to Change | 3, 6 and 9 weeks
  Motivation to Change will be assessed using University of Rhode Island Change Assessment (URICA). URICIA is a self report instrument that consists of 32 items. The range of scores is from 32 to 160, where a higher score indicates GREATER motivation to change.
Intimate Partner Violence (IPV) | Baseline and 9 Weeks
  IPV perpetration will be assessed using the Abusive Behavior Inventory (ABI). The ABI is a 30 item inventory that uses a 5 point Likert scale for each response. The greater the score, the greater the severity.
Substance Abuse | Baseline and 9 Weeks
  Substance abuse will be assessed using the Short-Michigan Alcohol Screening Test and the Drug Abuse Screening Test-10. This 10 item inventory characterizes behavior associated with alcoholism, the higher the score, the greater the severity of alcoholism in a respondent.
Parenting Behaviors | Baseline and 9 Weeks
  Parenting behaviors will be assessed with Parental Acceptance Rejection Questionnaire which includes 24 items on a 4 point likert scale. Higher scores mean greater negative parenting behaviors.
Co-Parenting Behaviors | Baseline and 9 Weeks
  Co-parenting behaviors will be assessed using the Coparenting Relationship Scale.
Perspective Taking | Baseline and 9 weeks
  The Perspective Taking Questionnaire is a 7 item questionnaire measured on a 5 point likert scale. Higher scores mean better perspective taking

CONTACTS AND LOCATIONS:
Locations (1):
- Yale University Child Study Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No